CLINICAL TRIAL: NCT00464854
Title: Feasiblity, Safety And Efficacy Of Glucose Control With Multiple Daily Insulin Injections In Diabetic Patients Hospitalized In A General Medicine Ward
Brief Title: Glucose Control With Multiple Daily Insulin Injections In Diabetic Patients Hospitalized In A General Medicine Ward
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was started before the official request for protocol registration
Sponsor: Assaf-Harofeh Medical Center (Other Government)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AH-2323
Record Dates: First submitted 2007-04-22; First posted 2007-04-24 (Estimated); Last update posted 2007-04-24 (Estimated); Status verified 2007-04

CONDITIONS: Diabetes Mellitus
Keywords: Glucose control; Subcutaneous insulin treatment; Multiple daily injections
MeSH Terms: conditions — Diabetes Mellitus | interventions — Insulin Glargine; Insulin Aspart; Insulin Lispro

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Glargine and insulin aspart or lispro

SUMMARY:
At least 20% of patients hospitalized in the general medical and surgical wards at any given time suffer from diabetes. It has been demonstrated that poor clinical outcome correlates with the degree of hyperglycemia in these patients. Strict glucose control in hospitalized patients improves clinical outcomes in the setting of acute myocardial infarction, cardiac surgical procedures, infection and critical illness in patients hospitalized in intensive care units if insulin is applied intravenously. It is, however, complex to obtain strict glucose control in the general surgical and medical wards. These wards are usually understaffed as compared to intensive care units and therefore are incapable to perform the necessary close monitoring essential in patients treated with intravenous insulin. We intend to test the feasibility of glucose control by multiple daily subcutaneous injections with long acting basal glargine insulin and pre-meal insulin analogues. If good glucose control can be achieved, this would be a valid, more convenient and acceptable alternative to intravenous insulin infusions to obtain good glucose control in diabetic patients hospitalized in general internal medicine wards.

DETAILED DESCRIPTION:
Location of the study:

Internal Medicine Wards C of Assaf Harofe Medical Center, Zerifin, Israel:

Inclusion Criteria:

* Adult (<18 years) Male and female T1 & T2DM patients who can sign an informed consent.
* Insulin treatment (at least one injection a day) prior to hospitalization for at least half a year.

Exclusion Criteria:

* Diabetic ketoacidosis.
* Hyperosmolar state due to hyperglycemia.
* Pregnancy
* Fertile women who do not use oral contraception or IUD

Concurrent medications:

· The hospital staff will determine the initiation or continuation of oral and intravenous medications as indicated by the patient's medical status.

Admission Blood tests:

* Routine: CBC, Creatinine, Urea, Na, K, GOT, GPT, Alp, Albumin, Glu
* HbA1C & Fructosamine.

Initiation and Titration of Insulin dosage:

* Glargine insulin will be initiated as a function of the first fasting glucose level and the patients body weight (0.3 - 0.8 U/kg). Up- or down titration will occur every morning by 10 - 20% according to capillary am fasting glucose (goal 130 mg%). The dosage of premeal insulin analogues will be based according to a sliding scale and calculated as a percentage of the amount of am glargine.
* Capillary blood glucose levels were measured seven times a day: before and two hours after breakfast, lunch and dinner and at bedtime. Additional measurements were performed according to clinical needs such as suspected hypoglycemia or unexplained deterioration of clinical condition

ELIGIBILITY:
Inclusion Criteria:

* Adult (<18 years) Male and female T1 & T2DM patients who can sign an informed consent.
* Insulin treatment (at least one injection a day) prior to hospitalization for at least half a year.

Exclusion Criteria:

* Diabetic ketoacidosis.
* Hyperosmolar state due to hyperglycemia.
* Pregnancy
* Fertile women who do not use oral contraception or IUD

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 2005-07; Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Achievement of a fasting blood glucose of 130 mg/dl and a mean daily glucose level of 180 mg/dl during hospitalization

SECONDARY OUTCOMES:
Hypoglycemia of < 60 mg% (symptomatic and asymptomatic)

CONTACTS AND LOCATIONS:
Overall Officials: Andreas E Buchs, M.D., Principal Investigator — Assaf Harofe Medical Center
Locations (1):
- Assaf Harofe Medical Center, Ẕerifin, Israel